CLINICAL TRIAL: NCT02163408
Title: 3D Multi-Contrast Atherosclerosis Characterization of the Carotid Artery
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Heart Association (Other)
Responsible Party: Principal Investigator, Debiao Li, PhD, Director, Biomedical Imaging Research Institute, Cedars-Sinai Medical Center
Other Study IDs: 35762; 2R01HL096119-05 (NIH)
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Carotid Artery Disease
Keywords: MRI; Plaque Characterization
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Volunteers: 100 healthy volunteers will take MRI with/without contrast using both conventional protocol and our developed protocol. Image quality and image contrast will be compared between the two protocols.
  Interventions: Other: MRI with/without contrast
- Patients with Carotid Artery Disease: 40 patients will take MRI with/without contrast using both conventional protocol and our developed protocol. Image quality, image contrast, and composition analysis will be compared between the protocols.

INTERVENTIONS:
Other: MRI with/without contrast — Bilateral carotid plaque imaging at 3.0T. Conventional MRI scans with T1-, T2-weightings and scans using the developed techniques. MR contrast may be used in conventional protocol when it is needed to evaluate the performance of the developed techniques
  Groups: Healthy Volunteers

SUMMARY:
This is a technical development study with the goal to develop 3D techniques for atherosclerosis plaque characterization. We hypothesize that 3D MRI is superior to 2D MRI in characterizing major plaque constituents that contribute to severe clinical events such as myocardial infarction or stroke. The major advantages of the 3D techniques to be developed will include high spatial resolution, reduced scan times, and optimized image contrast. The use of contrast injection is not needed with the new techniques, which is greatly beneficial for patients with advanced chronic kidney disease.This is not a funded clinical trial.

DETAILED DESCRIPTION:
All participants will undergo the conventional MRI protocol and the new imaging protocol using our developed techniques. They may have either non-contrast scans or contrast-enhanced scans or both depending on the stage of development. The comparison results between the two protocols will be used to evaluate the performance of the new techniques and help optimization of specific technical aspects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers: male or female ≥ 18 years of age with a BMI<30, with no history of cardiovascular disease
* Patients: Medically stable, male or female ≥ 18 years of age diagnosed with an atherosclerotic plaque in the carotid artery who have not undergone stenting of the carotid artery to be imaged.
* Ability to read and understand informed consent

Exclusion Criteria:

* Contraindications to MRI including mechanically, magnetically, or electrically activated implants, ferromagnetic implants and ferromagnetic foreign bodies, pregnancy.
* Inability to tolerate MRI secondary to an inability to lie supine or severe claustrophobia.
* Non-compliant with visit instructions, including inability to lie still, hold breath or follow procedure instructions
* Severe allergy to animal dander or animal-instigated asthma
* Specific to gadolinium-based contrast agents: Renal function test does not meet CSMC standard of care MRI contrast protocol requirements (GFR <45ml/min) or previous allergic reaction to gadolinium-based contrast agents.*

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 healthy volunteers and 40 patients with carotid artery disease will be recruited for this technical development study.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Image quality score | Within one year of scans
  Images collected from both investigational MRI pulse sequences and conventional protocol will be reviewed and scored by readers and compared.
Adverse plaque characteristics detection | Within one year of scans
  In patient study, the analysis of adverse plaque characteristics will be performed and compared between the conventional protocol and developed protocol.

SECONDARY OUTCOMES:
Image contrast-to-noise ratio | Within one year of scans
  Contrast-to-noise ratio will be measured on the images collected with the conventional protocol and developed protocol and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Debiao Li, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States